CLINICAL TRIAL: NCT07246356
Title: A Study to Explore the Feasibility and Efficacy of Group Traumatic Episode Protocol (GTEP) for Reducing Trauma Symptoms Following a Traumatic Birthing Experience
Brief Title: Feasibility and Efficacy of GTEP for Birth Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Black Country Healthcare NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_24-029; 341922 (Other: IRAS)
Record Dates: First submitted 2025-07-25; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: PTSD (Childbirth-Related); Psychological Wellbeing; Bonding
Keywords: GTEP; Group EMDR; Birth trauma; Psychological wellbeing; Perinatal; Parent infant bonding
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Birth Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GTEP (Experimental): Participants will receive the GTEP intervention, delivered online.
  Interventions: Behavioral: Group Traumatic Episode Protocol (GTEP)

INTERVENTIONS:
Behavioral: Group Traumatic Episode Protocol (GTEP) — GTEP is a group version of the Recent Traumatic Episode Protocol (R-TEP), a form of EMDR.
  The GTEP intervention will involve 2 sessions focusing on preparation (e.g., through grounding and emotional regulation) followed by 4 processing sessions.

SUMMARY:
This clinical study aims to evaluate the feasibility and initial efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms (measured by the PCL-5 and City BiTS) for individuals following a traumatic birthing experience. A secondary aim is to evaluate the efficacy of GTEP in improving parental wellbeing (measured through the CORE-10) and parent-infant bonding (measured through the PBQ) following a traumatic birthing experience.

Participants (those who have experienced a traumatic birthing experience) will complete the GTEP intervention, delivered online. They will be asked to complete outcome measures and give feedback on their experience of the group.

DETAILED DESCRIPTION:
It is estimated that up to 15.7% of individuals will experience some trauma symptoms following childbirth, with 4-6% developing Post-Traumatic Stress Disorder. Research has found there to be an increased risk of postpartum depression, postpartum psychosis and anxiety following a complicated or traumatic childbirth, along with reduced parent-infant bonding at 1, 6 and 12-months postpartum. Group Traumatic Episode Protocol (GTEP) is a version of Eye Movement Desensitization and Reprocessing (EMDR) to be used in group settings. There is a growing evidence base for the efficacy of GTEP in other populations and it has been found to reduce trauma symptoms in a refugee population, adult cancer patients and healthcare professionals . However, there is no research to date exploring the feasibility and efficacy of GTEP for trauma symptoms related to birth.

This study aims to evaluate the feasibility and efficacy of GTEP for reducing trauma symptoms (measured by the PCL-5 and City BiTS) for individuals following a traumatic birthing experience. Feasibility / acceptability will be evaluated using structured measures, along with open-ended qualitative questions. The facilitators of the group will also be administered these measures and asked for qualitative feedback about their experience of facilitating the group.

A secondary aim is to evaluate the efficacy of GTEP in improving parental wellbeing (measured through the CORE-10) and parent-infant bonding (measured through the PBQ) following a traumatic birthing experience

The GTEP Intervention (for use in this study):

The intervention will involve a total of 8 sessions:

* Session 1: a home visit to gain consent, determine full eligibility and complete outcome measures.
* Sessions 2 - 7: 6 online GTEP sessions, conducted via Zoom, which will happen weekly. Each session will last approximately 90 minutes.
* Session 8: A post-group follow-up, either face-to-face or over the telephone, to discuss experiences of the group, discuss any onward referrals (as required), complete final outcome measures.

Study Design:

This study will use a pre-post design, with outcome measure questionnaires (CORE-10, City BiTS, PBQ) completed at two time points (before and after the GTEP intervention). In addition, the primary outcome measure of the PCL-5, will be administered at 8 time points (i.e., during the pre-intervention home visit, before sessions 2, 3, 4, 5, 6 and 7 and during the post-intervention follow-up).

A study feasibility measure will also be administered to evaluate the feasibility of the intervention for this population. This will be administered to both client participants and the group facilitators, where appropriate. Qualitative feedback will also be gathered.

Participants:

Participants will be recruited via the Black Country Perinatal Mental Health Service (BCPMHS) who are self-reporting trauma symptoms related to a traumatic birthing experience within the last 18 months.

Data Analysis:

Data will be analysed at the University of Birmingham. Quantitative data analysis will include a pre-and-post-intervention comparison scores at both an individual (using a Reliable Change Index) and a group level (using either a bootstrapped paired samples t-test or a matched-pairs Wilcoxon). Descriptive statistics will also be used where appropriate.

Qualitative analysis may be conducted related to the feasibility questions outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years.
* Currently under the Black Country Perinatal Mental Health Service
* Experiencing self-reported trauma symptoms related to a birthing experience within the last 18 months (this includes the birth itself, the postnatal hospital stay, and/or any neonatal admissions).
* Access to technology (e.g., laptop, internet connection) to be able to access the online group.
* Access to a confidential space within their home, and childcare for their baby/any other existing children.
* Proficient levels of English Language to engage with the group.
* Ability to engage in group therapy based on clinical presentation.
* Capacity to consent to engage in the GTEP group and research study.

Exclusion Criteria:

* Pregnant people
* Women/birthing people whose baby is no longer under their care.
* Severe and enduring mental health presentations (i.e., diagnosis of bipolar, psychosis and/or schizophrenia.
* Significant sensory impairment (e.g., needing a British Sign Language interpreter).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | From enrolment to post-treatment follow-up session, from baseline up to 24 weeks.
  PCL-5 questionnaire to measure any changes in trauma symptoms. Scores can range between 0-80. The cut-off score for indicating probable PTSD is 31-33.

SECONDARY OUTCOMES:
City Birth Trauma Scale (CiBTS) | From enrolment through to post-intervention follow-up, from baseline up to 24 weeks.
  To measure trauma symptoms related directly to the childbirth experience. Scores on this measure range from 0-60, with higher scores indicating greater likelihood of trauma symptoms related to a childbirth experience.
Clinical Outcomes in Routine Evaluation 10 (CORE-10) | From enrolment through to post-intervention follow-up session, from baseline up to 24 weeks.
  A measure of psychological wellbeing. Scores range from 0-40, with higher scores indicating higher levels of distress. A score of 11 or above is generally considered clinically significant.
Parental Bonding Questionnaire (PBQ) | From enrolment through to post-intervention follow-up session, from baseline up to 24 weeks.
  To measure levels of parent-infant bonding. Scores can range from 0-125, with higher scores indicating greater bonding difficulties.
Acceptability of Intervention Measure (AIM) | From session 2 to post-treatment follow up session, up to 24 weeks.
  These measured are used to help evaluate the feasibility and acceptability of the GTEP intervention. These questions will be asked at the beginning of each session from T2 - T8. Questionnaires have been based on these measures but adapted for this specific population. Scores can range from 13-70, with higher scores indicating greater acceptability / feasibility.
Feasibility of Intervention Measure (FIM) | From session 2 to post-treatment follow up session, up to 24 weeks.
  This measure is used to help evaluate the feasibility of the G-TEP intervention. Questionnaires have been based on these measures but adapted for this specific population. Scores can range from 13-70, with higher scores indicating greater acceptability / feasibility. These questions will be asked at the beginning of each session from T2 - T8.
Intervention Appropriateness Measure (IAM) | From session 2 to post-treatment follow up session, up to 24 weeks.
  This measure is used to help evaluate the appropriateness of the G-TEP intervention for this population group. These questions will be asked at the beginning of each session from T2 - T8. Questionnaires have been based on these measures but adapted for this specific population. Scores can range from 13-70, with higher scores indicating greater acceptability / feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Strachan, Study Principal Investigator, Principal Investigator — Black Country Healthcare NHS Foundation Trust; Alice Welham, Study Co-Investigator, Study Chair — University of Birmingham
Locations (1):
- Black Country Healthcare NHS Foundation Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ertan D, Hingray C, Burlacu E, Sterle A, El-Hage W. Post-traumatic stress disorder following childbirth. BMC Psychiatry. 2021 Mar 16;21(1):155. doi: 10.1186/s12888-021-03158-6. PMID 33726703
- [Background] Kjerulff KH, Attanasio LB, Sznajder KK, Brubaker LH. A prospective cohort study of post-traumatic stress disorder and maternal-infant bonding after first childbirth. J Psychosom Res. 2021 May;144:110424. doi: 10.1016/j.jpsychores.2021.110424. Epub 2021 Mar 17. PMID 33756149
- [Background] Yurtsever A, Konuk E, Akyuz T, Zat Z, Tukel F, Cetinkaya M, Savran C, Shapiro E. An Eye Movement Desensitization and Reprocessing (EMDR) Group Intervention for Syrian Refugees With Post-traumatic Stress Symptoms: Results of a Randomized Controlled Trial. Front Psychol. 2018 Jun 12;9:493. doi: 10.3389/fpsyg.2018.00493. eCollection 2018. PMID 29946275
- [Background] Roberts, A. K. P. (2018). The effects of the EMDR group traumatic episode protocol with cancer survivors. Journal of EMDR Practice and Research, 12(3), 105-117. https://doi.org/10.1891/1933-3196.12.3.105
- [Background] Tsouvelas, G., Chondrokouki, M., Nikolaidis, G., & Shapiro, E. (2019). A vicarious trauma preventive approach. The Group Traumatic Episode Protocol EMDR and workplace affect in professionals who work with child abuse and neglect. 2, 130-138. https://doi.org/10.26386/obrela.v2i3.123
- [Background] Farrell D, Moran J, Zat Z, Miller PW, Knibbs L, Papanikolopoulos P, Prattos T, McGowan I, McLaughlin D, Barron I, Matthess C, Kiernan MD. Group early intervention eye movement desensitization and reprocessing therapy as a video-conference psychotherapy with frontline/emergency workers in response to the COVID-19 pandemic in the treatment of post-traumatic stress disorder and moral injury-An RCT study. Front Psychol. 2023 Mar 23;14:1129912. doi: 10.3389/fpsyg.2023.1129912. eCollection 2023. PMID 37063579
- [Background] Pink, J., Ghomi, M., Smart, T., & Richardson, T. (2022). Effects of EMDR Group Traumatic Episode Protocol on Burnout Within IAPT Healthcare Professionals: A Feasibility and Acceptability Study. Journal of EMDR Practice and Research, 16(4), 215-227. https://doi.org/10.1891/EMDR-2022-0029
- [Background] Barkham, M., Bewick, B., Mullin, T., Gilbody, S., Connell, J., Cahill, J., Mellor-Clark, J., Richards, D., Unsworth, G., & Evans, C. (2013). The CORE-10: A short measure of psychological distress for routine use in the psychological therapies. Counselling and Psychotherapy Research, 13, 3-13. https://doi.org/10.1080/14733145.2012.729069
- [Background] Brockington, I. F., Oates, J., George, S., Turner, D., Vostanis, P., Sullivan, M., Loh, C., & Murdoch, C. (2001). A Screening Questionnaire for mother-infant bonding disorders. Archives of Women's Mental Health, 3(4), 133-140. https://doi.org/10.1007/s007370170010
- [Background] Ayers S, Wright DB, Thornton A. Development of a Measure of Postpartum PTSD: The City Birth Trauma Scale. Front Psychiatry. 2018 Sep 18;9:409. doi: 10.3389/fpsyt.2018.00409. eCollection 2018. PMID 30279664
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Shapiro, E (2013). "The EMDR Group Traumatic Episode Protocol." Presentation to the EMDR Turkey Conference, Istanbul, Turkey.
- [Background] Shapiro, E., & Laub, B. (2008). Early EMDR Intervention (EEI): A Summary, a Theoretical Model, and the Recent Traumatic Episode Protocol (R-TEP). Journal of EMDR Practice and Research, 2(2), 79-96. https://doi.org/10.1891/1933-3196.2.2.79
- See also: PTSD UK — https://www.ptsduk.org

DOCUMENTS (3):
  • Study Protocol (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT07246356/Prot_000.pdf
  • Informed Consent Form: Facilitator consent form (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT07246356/ICF_001.pdf
  • Informed Consent Form: Participant consent form (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT07246356/ICF_002.pdf